CLINICAL TRIAL: NCT02540265
Title: A Phase 2, Single-Center, Randomized, Double-Blind, Placebo-Controlled, Evaluation of the Safety, Efficacy, and Pharmacokinetics of N1539 Following Bunionectomy
Brief Title: Placebo-Controlled Evaluation of N1539 Following Bunionectomy Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baudax Bio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REC-15-014
Record Dates: First submitted 2015-08-31; First posted 2015-09-03 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Pain, Post-operative
Keywords: Bunion; Bunionectomy; Pain; Analgesia; N1539
MeSH Terms: conditions — Pain, Postoperative; Bunion; Pain; Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- N1539 30mg (Experimental): N1539 (Intravenous meloxicam) 30mg every 24 hours for up to 3 doses.
  Interventions: Drug: N1539
- N1539 60mg (Experimental): N1539 (Intravenous meloxicam) 60mg every 24 hours for up to 3 doses.
  Interventions: Drug: N1539
- IV Placebo (Placebo Comparator): IV Placebo every 24 hours for up to 3 doses.
  Interventions: Drug: Intravenous Placebo

INTERVENTIONS:
Drug: N1539
  Other Names: Intravenous meloxicam
  Arms: N1539 30mg; N1539 60mg
Drug: Intravenous Placebo
  Arms: IV Placebo

SUMMARY:
The primary objective of this study is to evaluate the safety of N1539 in subjects with acute moderate to severe pain following unilateral bunionectomy.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily provide written informed consent.
* Male or female between 18 and 75 years of age, inclusive.
* Be scheduled to undergo a primary unilateral first metatarsal bunionectomy repair
* Be American Society of Anesthesiology (ASA) physical class 1 or 2.
* Female subject are eligible only if all the following apply:

  * Not pregnant;
  * Not lactating;
  * Not planning to become pregnant during the study;
  * Commit to the use of an acceptable form of birth control for the duration of the study through Day 30.
* Have a body mass index ≤35 kg/m2
* Be able to understand the study procedures, comply with all study procedures, and agree to participate in the study program.

Exclusion Criteria:

* Have a known allergy to meloxicam or any excipient of N1539, D5W, aspirin, other non-steroidal anti-inflammatory drugs (NSAIDs) or to any peri- or postoperative medications used in this study.
* Have a clinically significant abnormal clinical laboratory test value.
* Have history of or positive test results for HIV, or hepatitis B or C.
* Have a history or clinical manifestations of significant renal, hepatic, cardiovascular, metabolic, neurologic, psychiatric, or other condition that would preclude participation in the study.
* Have a history of migraine or frequent headaches, seizures, or are currently taking anticonvulsants.
* Have another painful physical condition that may confound the assessments of post operative pain.
* Have a history of syncope or other syncopal attacks.
* Have evidence of a clinically significant 12 lead ECG abnormality.
* Have a history of alcohol abuse (regularly drinks > 4 units of alcohol per day; 8 oz. beer, 3 oz. wine, 1 oz. spirits) or prescription/illicit drug abuse..
* Have positive results on the urine drug screen or alcohol breath test indicative of illicit drug or alcohol abuse.
* Have been receiving or have received chronic opioid therapy defined as greater than 15 morphine equivalents units per day for greater than 3 out of 7 days per week over a one-month period within 12 months.
* Use concurrent therapy that could interfere with the evaluation of efficacy or safety, such as any drugs which in the investigator's opinion may exert significant analgesic properties or act synergistically with N1539.
* Unable to discontinue medications, that have not been at a stable dose for at least 14 days prior to the scheduled bunionectomy procedure, within 5 half lives of the specific prior medication (or, if half life is not known, within 48 hours) before dosing.
* Have utilized corticosteroids, either systemically, inhalational either intranasally or oral, or by intra-articular injection, within 14 days prior to the study.
* Have received any investigational product within 30 days before dosing with study medication.
* Be receiving warfarin, lithium, or a combination of furosemide with either an angiotensin converting enzyme inhibitor or an angiotensin receptor blocker
* Be currently receiving treatment with oral meloxicam (Mobic®)
* Have previously received N1539 in clinical trials, or had bunionectomy in the last 3 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2015-08; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Chesapeake Research Group, LLC, Pasadena, Maryland, United States

REFERENCES:
- [Derived] Viscusi ER, Gan TJ, Bergese S, Singla N, Mack RJ, McCallum SW, Du W, Hobson S. Intravenous meloxicam for the treatment of moderate to severe acute pain: a pooled analysis of safety and opioid-reducing effects. Reg Anesth Pain Med. 2019 Mar;44(3):360-368. doi: 10.1136/rapm-2018-100184. Epub 2019 Feb 7. PMID 30737315

RESULTS

PARTICIPANT FLOW:
Groups:
- N1539 30mg: N1539 (Intravenous meloxicam) 30mg every 24 hours for up to 3 doses.
  N1539
- N1539 60mg: N1539 (Intravenous meloxicam) 60mg every 24 hours for up to 3 doses.
  N1539
- IV Placebo: IV Placebo every 24 hours for up to 3 doses.
  Intravenous Placebo
Period: Overall Study
Arm/Group | N1539 30mg | N1539 60mg | IV Placebo
Started | 20 | 20 | 19
Treatment Completion (Subjects receiving at least 2 study doses were considered as treatment complete) | 20 | 19 | 18
Completed (Subjects who completed the final study followup were considered study completers) | 20 | 20 | 18
Not Completed | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Analysis population includes all subjects randomized to treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | N1539 30mg | N1539 60mg | IV Placebo | Total
Number analyzed (Participants) | 20 | 20 | 19 | 59
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1 | 2
  Between 18 and 65 years | 19 | 16 | 16 | 51
  >=65 years | 1 | 3 | 2 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.6 (12.66) | 44.9 (16.67) | 49.2 (12.81) | 47.2 (14.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 18 | 14 | 48
  Male | 4 | 2 | 5 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 0 | 3
  Not Hispanic or Latino | 17 | 20 | 19 | 56
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 10 | 9 | 11 | 30
  White | 10 | 10 | 8 | 28
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 19 | 59
Baseline Pain Intensity (0-10 NPRS) [Mean (Standard Deviation); unit: units on a scale] — Pain intensity was recorded using a Numeric Pain Rating Scale (NPRS; Range 0-10) where 0 equates to no pain (better), and 10 equates to the worst pain imaginable (worse).
  units on a scale | 7.7 (2.00) | 7.4 (1.90) | 7.7 (2.24) | 7.6 (2.02)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Adverse Events
Description: Number of subjects reporting treatment emergent adverse events
Time Frame: Through Day 30 Follow-up
Population: All subjects treated with ≥1 dose of study medication (Safety analysis set)
Measure: Count of Participants; unit: Participants
Arm/Group | N1539 30mg | N1539 60mg | IV Placebo
Number analyzed (Participants) | 20 | 20 | 19
Participants | 12 | 10 | 10

2. Secondary Outcome: Effect Size of N1539 Doses Using the Summed Pain Intensity Difference Over the First 48 Hours (SPID48)
Description: Effect size was estimated based on SPID48 derived using 2-hour windowed last observation carried forward (W2LOCF) method and an analysis of covariance (ANCOVA) model that included treatment and baseline PI score.
Time Frame: 48 Hours
Population: All subjects treated with ≥1 dose of study medication and who had baseline PI and at least one post baseline PI (mITT analysis set; efficacy analysis set)
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | N1539 30mg | N1539 60mg | IV Placebo
Number analyzed (Participants) | 20 | 20 | 19
units on a scale | -9241.9 (1411.74) | -8350.6 (1413.30) | -1991.3 (1448.20)
Statistical Analysis 1: Comparison: N1539 30mg vs IV Placebo; Test type: Other; Effect Size = 1.01
Statistical Analysis 2: Comparison: N1539 60mg vs IV Placebo; Test type: Other; Effect Size = 0.87

3. Secondary Outcome: Summed Pain Intensity Difference Over the First 48 Hours (SPID48)
Description: Pain intensity was recorded using a Numeric Pain Rating Scale (Range 0-10) where 0 equates to no pain (better), and 10 equates to the worst pain imaginable (worse). Pain intensity scores were to be recorded at the following time points: 0.25, 0.5, 0.75, 1, 2, 4, and 6 hours post Dose 1. Thereafter pain assessments were to be recorded every 2 hours until 48 hours post Dose 1. Pain intensity differences from baseline at each time point were calculated and a time weighted summed pain intensity difference (SPID) was then calculated. Time weighted SPID calculations were computed by multiplying a weight factor to each score prior to summation. The weight factor at each time point was the time elapsed since the previous observation. A smaller SPID was better.
Time Frame: 48 Hours
Population: mITT analysis set
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | N1539 30mg | N1539 60mg | IV Placebo
Number analyzed (Participants) | 20 | 20 | 19
units on a scale | -9241.9 (1411.74) | -8350.6 (1413.30) | -1991.3 (1448.20)
Statistical Analysis 1: Comparison: N1539 30mg vs IV Placebo; Test type: Superiority; p = 0.0049, t-test, 2 sided
Statistical Analysis 2: Comparison: N1539 60mg vs IV Placebo; Test type: Superiority; p = 0.0076, t-test, 2 sided

4. Secondary Outcome: Summed Pain Intensity Difference (SPID) at Other Intervals
Description: as for outcome 3
Time Frame: 48 Hours
Population: mITT analysis set
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | N1539 30mg | N1539 60mg | IV Placebo
Number analyzed (Participants) | 20 | 20 | 19
units on a scale
  SPID6 (Hour 0-6) | -793.87 (172.45) | -663.17 (172.64) | 146.22 (176.91)
  SPID12 (Hour 0-12) | -1655.1 (338.78) | -1334.9 (339.15) | 319.67 (347.53)
  SPID24 (Hour 0-24) | -3024.0 (644.63) | -2793.3 (645.34) | 276.46 (661.28)
  SPID12-24 (Hour 12-24) | -1368.9 (343.34) | -1458.4 (343.72) | -43.21 (352.21)
  SPID12-48 (Hour 12-48) | -7586.8 (1121.12) | -7015.7 (1122.35) | -2311.0 (1150.07)
  SPID24-48 (Hour 24-48) | -6217.9 (817.22) | -5557.3 (818.12) | -2267.8 (838.33)
Statistical Analysis 1: Comparison: N1539 30mg vs IV Placebo; Test type: Superiority; p < 0.05, t-test, 2 sided — Applies to SPID 0-6, SPID 0-12, SPID 0-24, SPID 12-24, SPID 12-48, and SPID 24-48
Statistical Analysis 2: Comparison: N1539 60mg vs IV Placebo; Test type: Superiority; p < 0.05, t-test, 2 sided — Applies to SPID 0-6, SPID 0-12, SPID 0-24, SPID 12-24, SPID 12-48, and SPID 24-48

5. Secondary Outcome: Number of Subjects With Use of Rescue Medication (Oral Opioids)
Time Frame: 48 hours
Population: mITT analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | N1539 30mg | N1539 60mg | IV Placebo
Number analyzed (Participants) | 20 | 20 | 19
Participants
  Hour 0-24 | 20 | 18 | 19
  Hour 24-48 | 11 | 10 | 14
  Hour 0-48 | 20 | 18 | 19

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | N1539 30mg | N1539 60mg | IV Placebo
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/19
Other Adverse Events (participants affected / at risk) | 12/20 | 10/20 | 10/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | N1539 30mg (N=20) | N1539 60mg (N=20) | IV Placebo (N=19)
Nausea (Gastrointestinal disorders) | 6 (9) | 4 (5) | 4 (8)
Headache (Nervous system disorders) | 2 (2) | 3 (5) | 4 (8)
Dizziness (Nervous system disorders) | 3 (6) | 2 (2) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2) | 2 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (4) | 0 (0) | 1 (2)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Discussion and/or publication of data generated is not permitted without the prior written consent of the sponsor.